CLINICAL TRIAL: NCT00234832
Title: Sibutramine Cardiovascular Morbidity/Mortality Outcomes Study in Overweight or Obese Subjects at Risk of a Cardiovascular Event
Brief Title: A Long Term Study of Sibutramine and the Role of Obesity Management in Relation to Cardiovascular Disease in Overweight and Obese Patients
Acronym: SCOUT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Cheryl Renz, MD, Abbott
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M01-392
Record Dates: First submitted 2005-09-13; First posted 2005-10-10 (Estimated); Results first posted 2010-04-15 (Estimated); Last update posted 2010-05-11 (Estimated); Status verified 2010-05

CONDITIONS: Obesity
Keywords: Obesity; Sibutramine
MeSH Terms: conditions — Obesity | interventions — sibutramine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Sibutramine (Experimental): Subjects were randomized to receive sibutramine 10 mg once daily (QD) during the Treatment Period after a 6-week Lead-in Period
  Interventions: Drug: Sibutramine hydrochloride
- Placebo (Placebo Comparator): Subjects were randomized to receive placebo QD during the Treatment Period after a 6-week Lead-in Period
  Interventions: Drug: Placebo
- Lead-in sibutramine (Experimental): All subjects received 10 mg sibutramine QD during a 6-week Lead-in Period
  Interventions: Drug: Sibutramine hydrochloride

INTERVENTIONS:
Drug: Sibutramine hydrochloride — One 10 mg tablet QD plus country-specific standard care for weight management. (During the Treatment Period, the dose could have been titrated up to 15 mg at the investigator's discretion.)
  Other Names: ABT-991; sibutramine; Meridia; Reductil
  Arms: Sibutramine
Drug: Placebo — 1 tablet QD plus country-specific standard care for weight management (During the Treatment Period, the dose could have been titrated up to 15 mg at the investigator's discretion.)
  Arms: Placebo
Drug: Sibutramine hydrochloride — 10 mg tablet QD during the 6-week Lead-in Period plus country-specific standard care for weight management
  Arms: Lead-in sibutramine

SUMMARY:
The purpose of the study was to determine the long-term effect of sibutramine treatment on cardiovascular outcomes in overweight and obese patients at risk of a cardiovascular event.

DETAILED DESCRIPTION:
The study consisted of 4 periods: 1) a Screening Period of approximately 2 weeks; 2) a 6-week Lead-in Period, during which subjects received single-blind sibutramine and country-specific standard of care for weight management. Subjects who discontinued study drug treatment during the Lead-in Period were not randomized and did not participate in the double-blind Treatment Period or the Follow-up Period; 3) a double-blind Treatment Period in which subjects were randomized to 1 of the 2 treatment groups and were followed until the study ended; and 4) a double-blind Follow-up Period, during which randomized subjects who discontinued study drug were followed until the study ended. The Randomization Phase consisted of the double-blind Treatment Period and the double-blind Follow-up Period. Subjects received country-specific standard of care for weight management during the Randomization Phase.

An independent events adjudication committee evaluated all potential cardiovascular outcome events and confirmed the outcome events and time of onset to be included in the statistical analyses.

ELIGIBILITY:
Inclusion Criteria:

* Subject's body mass index (BMI) was >= 27 kg/m(2) and <= 45 kg/m(2) or their BMI was >= 25 kg/m(2) and < 27 kg/m(2) with waist circumference of >= 102 cm in males or >= 88 cm in females.
* Medical history positive for:

  * Preexisting cardiovascular disease (i.e., coronary artery disease, cerebrovascular disease, or peripheral arterial occlusive disease) and/or
  * Type 2 diabetes mellitus with at least 1 other risk factor (i.e., dyslipidemia, controlled hypertension, current smoker, or diabetic nephropathy with evidence of microalbuminuria)

Exclusion Criteria:

* History of recent myocardial infarction.
* Heart failure symptoms greater than New York Heart Association Functional Class II.
* Hemodynamically significant valvular or left ventricular (LV) tract obstruction.
* Subjects without a pacemaker and with any of the following:

  * Sinus bradycardia (< 50 bpm)
  * Sick sinus syndrome
  * Atrioventricular block of more than 1st degree
* Mean sitting systolic blood pressure (SBP) > 160 mmHg. Mean sitting diastolic blood pressure (DBP) > 100 mmHg. Mean sitting heart rate (HR) > 100 bpm.
* Syncopal episodes presumed to be due to uncontrolled life-threatening arrhythmias.
* Planned cardiac surgery or coronary angioplasty within 6 months of screening.
* History of recent non-hemorrhagic stroke or transient ischemic attack (TIA), history of hemorrhagic stroke.
* Hyperthyroidism.
* Known chronic liver disease or endstage renal disease.
* Severe, symptomatic benign prostatic hyperplasia which may require surgery.
* Known pheochromocytoma, history of narrow angle glaucoma, Gilles de la Tourette syndrome, history of seizures, history of bariatric or abdominal obesity surgery (excluding liposuction).
* Concomitant use of monoamine oxidase inhibitors or drugs that increase levels of serotonin in the brain.
* Treated hypertension stabilized for less than 3 months.
* Inability to perform regular physical activity.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10777 (Actual)
Dates: Start 2003-01; Primary Completion 2009-03 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl Renz, MD, Study Director — Abbott
Locations (1):
- Global Medical Services, North Chicago, Illinois, United States

REFERENCES:
- [Derived] Jorgensen ME, Torp-Pedersen C, Finer N, Caterson I, James WP, Legler UF, Andersson C. Association between serum bilirubin and cardiovascular disease in an overweight high risk population from the SCOUT trial. Nutr Metab Cardiovasc Dis. 2014 Jun;24(6):656-62. doi: 10.1016/j.numecd.2013.12.009. Epub 2014 Jan 18. PMID 24534073
- [Derived] Seimon RV, Espinoza D, Ivers L, Gebski V, Finer N, Legler UF, Sharma AM, James WP, Coutinho W, Caterson ID. Changes in body weight and blood pressure: paradoxical outcome events in overweight and obese subjects with cardiovascular disease. Int J Obes (Lond). 2014 Sep;38(9):1165-71. doi: 10.1038/ijo.2014.2. Epub 2014 Jan 10. PMID 24406481
- [Derived] James WP, Caterson ID, Coutinho W, Finer N, Van Gaal LF, Maggioni AP, Torp-Pedersen C, Sharma AM, Shepherd GM, Rode RA, Renz CL; SCOUT Investigators. Effect of sibutramine on cardiovascular outcomes in overweight and obese subjects. N Engl J Med. 2010 Sep 2;363(10):905-17. doi: 10.1056/NEJMoa1003114. PMID 20818901
- [Derived] Weeke P, Andersson C, Fosbol EL, Brendorp B, Kober L, Sharma AM, Finer N, James PT, Caterson ID, Rode RA, Torp-Pedersen C. The weight lowering effect of sibutramine and its impact on serum lipids in cardiovascular high risk patients with and without type 2 diabetes mellitus - an analysis from the SCOUT lead-in period. BMC Endocr Disord. 2010 Feb 26;10:3. doi: 10.1186/1472-6823-10-3. PMID 20184783
- [Derived] Andersson C, Weeke P, Brendorp B, Kober L, Fosbol EL, Sharma AM, Finer N, Caterson ID, Rode RA, James PT, Torp-Pedersen C. Differential changes in serum uric acid concentrations in sibutramine promoted weight loss in diabetes: results from four weeks of the lead-in period of the SCOUT trial. Nutr Metab (Lond). 2009 Oct 14;6:42. doi: 10.1186/1743-7075-6-42. PMID 19828038

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 10777 subjects enrolled into the study, 33 were not treated with Lead-in Period sibutramine. Of the 10744 subjects who took at least 1 dose of Lead-in Period sibutramine, 939 were not randomized. One of the remaining 9805 subjects was not dispensed randomized study drug and was not included in the intent-to-treat population (N = 9804).
Groups:
- Randomized Sibutramine: Subjects who completed the 6-week Lead-in Period and who were randomized and dispensed sibutramine during the Treatment Period and continued standard care for weight management. If sibutramine was prematurely discontinued, subjects continued standard care for weight management during the Follow-up Period.
- Randomized Placebo: Subjects who completed the 6-week Lead-in Period and who were randomized and dispensed placebo during the Treatment Period and continued standard care for weight management. If placebo was prematurely discontinued, subjects continued standard care for weight management during the Follow-up Period.
Period: Overall Study
Arm/Group | Randomized Sibutramine | Randomized Placebo
Started | 4906 (Subjects completed the 6-week Lead-in Period and were dispensed randomized study drug.) | 4898 (Subjects completed the 6-week Lead-in Period and were dispensed randomized study drug.)
Completed | 3890 (Subjects completed the Randomization Phase.) | 3902 (Subjects completed the Randomization Phase.)
Not Completed | 1016 | 996

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Randomized Sibutramine | Randomized Placebo | Total
Number analyzed (Participants) | 4906 | 4898 | 9804
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3040 | 2997 | 6037
  >=65 years | 1866 | 1901 | 3767
Age Continuous [Mean (Standard Deviation); unit: years] | 63.2 (6.09) | 63.3 (6.15) | 63.2 (6.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2099 | 2055 | 4154
  Male | 2807 | 2843 | 5650
Region of Enrollment [Number; unit: participants]
  Europe | 4160 | 4150 | 8310
  Australia | 384 | 385 | 769
  Brazil | 233 | 234 | 467
  Mexico | 129 | 129 | 258
Cardiovascular (CV) risk group status [Number; unit: Participants] — Subjects were categorized at study entry into 1 of 3 prespecified CV risk groups: 1) diabetes mellitus (DM) only = history of type 2 DM with at least one other risk factor but no history of CV disease, 2) CV only = history of coronary artery disease, cerebrovascular disease, or peripheral arterial occlusive disease, but no history of type 2 DM with at least one other risk factor, and 3) CV + DM = history of coronary artery disease, cerebrovascular disease, or peripheral arterial occlusive disease, and a history of type 2 DM with at least one other risk factor.
  Participants
    DM only | 1207 | 1178 | 2385
    CV only | 759 | 793 | 1552
    CV + DM | 2906 | 2901 | 5807
    Unknown CV risk group status | 34 | 26 | 60

OUTCOME MEASURES:

1. Primary Outcome: Risk of Experiencing a Primary Outcome Event (POE) (i.e., Nonfatal Myocardial Infarction [MI], Nonfatal Stroke, Resuscitated Cardiac Arrest, Cardiovascular [CV] Death)
Description: For each subject, POE status (with/without an event) and time to first occurrence of a POE using time-to-event analysis were evaluated. All POE confirmed by an independent adjudication committee were included in the analysis.
Time Frame: From randomization up to 6 years
Population: Analysis based on intent-to-treat (ITT) population, which consists of all randomized subjects dispensed randomized study drug and grouped according to the intervention to which they were randomized. Subjects were also categorized into 1 of 3 prespecified CV risk groups: diabetes mellitus (DM) only, CV only, and CV + DM.
Measure: Number; unit: Participants
Groups:
- DM Only Randomized to Sibutramine: Subjects with a history of type 2 DM with at least one other risk factor (i.e., hypertension controlled on medication, dyslipidemia, current cigarette smoking, diabetic nephropathy with evidence of microalbuminuria), but no history of coronary artery disease, cerebrovascular disease, or peripheral arterial occlusive disease who completed the 6-week Lead-in Period and who were randomized and dispensed sibutramine during the Treatment Period and continued standard care for weight management.
- DM Only Randomized to Placebo: Subjects with a history of type 2 DM with at least one other risk factor (i.e., hypertension controlled on medication, dyslipidemia, current cigarette smoking, diabetic nephropathy with evidence of microalbuminuria), but no history of coronary artery disease, cerebrovascular disease, or peripheral arterial occlusive disease who completed the 6-week Lead-in Period and who were randomized and dispensed placebo during the Treatment Period and continued standard care for weight management.
- CV Only Randomized to Sibutramine: Subjects with a history of coronary artery disease, cerebrovascular disease, or peripheral arterial occlusive disease, but no history of type 2 DM with at least one other risk factor who completed the 6-week Lead-in Period and who were randomized and dispensed sibutramine during the Treatment Period and continued standard care for weight management.
- CV Only Randomized to Placebo: Subjects with a history of coronary artery disease, cerebrovascular disease, or peripheral arterial occlusive disease, but no history of type 2 DM with at least one other risk factor who completed the 6-week Lead-in Period and who were randomized and dispensed placebo during the Treatment Period and continued standard care for weight management.
- CV + DM Randomized to Sibutramine: Subjects with a history of coronary artery disease, cerebrovascular disease, or peripheral arterial occlusive disease, and with a history of type 2 DM with at least one other risk factor who completed the 6-week Lead-in Period and who were randomized and dispensed sibutramine during the Treatment Period and continued standard care for weight management.
- CV + DM Randomized to Placebo: Subjects with a history of coronary artery disease, cerebrovascular disease, or peripheral arterial occlusive disease, and with a history of type 2 DM with at least one other risk factor who completed the 6-week Lead-in Period and who were randomized and dispensed placebo during the Treatment Period and continued standard care for weight management.
Arm/Group | Randomized Sibutramine | Randomized Placebo | DM Only Randomized to Sibutramine | DM Only Randomized to Placebo | CV Only Randomized to Sibutramine | CV Only Randomized to Placebo | CV + DM Randomized to Sibutramine | CV + DM Randomized to Placebo
Number analyzed (Participants) | 4906 | 4898 | 1207 | 1178 | 759 | 793 | 2906 | 2901
Participants
  Intent-to-treat population | 561 | 490 | 79 | 77 | 77 | 66 | 403 | 346
Statistical Analysis 1: Comparison: Randomized Sibutramine vs Randomized Placebo; For the sample size calculation, a two-tailed alpha level of 0.05 was used along with power of 90%. The annual composite event rate in the placebo arm was assumed to be 7.0%. A sample of 3983 subjects in each of the 2 groups, corrected for a 30% noncompliance rate (15% in Year 1 and 6.3% in each year, Years 2 to 4), followed for at least 3 years was expected to have 90% power to detect a relative risk reduction of 15% with sibutramine relative to placebo; Test type: Superiority or Other; p = 0.015, Log Rank — No adjustment for multiple testing or interim analysis was performed. The primary outcome was tested at a 2-sided alpha level of 0.05; Cox Proportional Hazard = 1.162, 95% CI 2-sided [1.029 to 1.311] — The Cox model included factors for treatment, country, gender, and age (continuous) at Lead-in Period baseline. For the calculation of risk, the sibutramine arm is the numerator and the placebo arm is the denominator
Statistical Analysis 2: Comparison: DM Only Randomized to Sibutramine vs DM Only Randomized to Placebo; This analysis included only subjects with DM only in a comparison of sibutramine and placebo; Test type: Superiority or Other; p = 0.948, Log Rank; Cox Proportional Hazard = 1.010, 95% CI 2-sided [0.738 to 1.384]
Statistical Analysis 3: Comparison: CV Only Randomized to Sibutramine vs CV Only Randomized to Placebo; This analysis included only subjects with CV only in a comparison of sibutramine and placebo; Test type: Superiority or Other; p = 0.149, Log Rank; Cox Proportional Hazard = 1.276, 95% CI 2-sided [0.916 to 1.776]
Statistical Analysis 4: Comparison: CV + DM Randomized to Sibutramine vs CV + DM Randomized to Placebo; This analysis included only subjects with CV + DM in a comparison of sibutramine and placebo; Test type: Superiority or Other; p = 0.022, Log Rank; Cox Proportional Hazard = 1.182, 95% CI 2-sided [1.024 to 1.365]

2. Secondary Outcome: Risk of Death From Any Cause (All-cause Mortality)
Description: For each subject who died, the time to death was evaluated using time-to-event analysis.
Time Frame: From randomization up to 6 years
Population: Analysis based on ITT population, which consists of all randomized subjects dispensed randomized study drug and grouped according to the intervention to which they were randomized.
Measure: Number; unit: Participants
Arm/Group | Randomized Sibutramine | Randomized Placebo
Number analyzed (Participants) | 4906 | 4898
Participants | 418 | 404
Statistical Analysis 1: Comparison: Randomized Sibutramine vs Randomized Placebo; Test type: Superiority or Other; p = 0.543, Log Rank; Cox Proportional Hazard = 1.043, 95% CI 2-sided [0.910 to 1.196]

3. Secondary Outcome: Risk of Experiencing a POE or a Revascularization Procedure
Description: This outcome includes nonfatal MI, nonfatal stroke, resuscitated cardiac arrest, CV death (including events such as fatal MI and fatal stroke), and any of the following revascularization procedures: percutaneous transluminal coronary angioplasty, coronary artery bypass graft, coronary artery stent placement, cardiac transplant, peripheral vascular bypass or angioplasty, and carotid endarterectomy. For each subject, the POE or revascularization status (yes/no) and time to first occurrence of an event using time-to-event analysis were evaluated.
Time Frame: From randomization up to 6 years
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Randomized Sibutramine | Randomized Placebo
Number analyzed (Participants) | 4906 | 4898
Participants | 927 | 856
Statistical Analysis 1: Comparison: Randomized Sibutramine vs Randomized Placebo; Test type: Superiority or Other; p = 0.051, Log Rank; Cox Proportional Hazard = 1.097, 95% CI 2-sided [0.999 to 1.204]

4. Secondary Outcome: Risk of Experiencing a Nonfatal MI Included in the POE
Description: For each subject, the first occurrence of a nonfatal MI included in the POE was evaluated using time-to-event analysis.
Time Frame: From randomization up to 6 years
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Randomized Sibutramine | Randomized Placebo
Number analyzed (Participants) | 4906 | 4898
Participants | 200 | 159
Statistical Analysis 1: Comparison: Randomized Sibutramine vs Randomized Placebo; Test type: Superiority or Other; p = 0.022, Log Rank; Cox Proportional Hazard = 1.276, 95% CI 2-sided [1.036 to 1.571]

5. Secondary Outcome: Risk of Experiencing a Nonfatal Stroke Included in the POE
Description: For each subject, the time to first occurrence of a nonfatal stroke included in the POE was evaluated using time-to-event analysis.
Time Frame: From randomization up to 6 years
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Randomized Sibutramine | Randomized Placebo
Number analyzed (Participants) | 4906 | 4898
Participants | 127 | 95
Statistical Analysis 1: Comparison: Randomized Sibutramine vs Randomized Placebo; Test type: Superiority or Other; p = 0.025, Log Rank; Cox Proportional Hazard = 1.355, 95% CI 2-sided [1.038 to 1.767]

6. Secondary Outcome: Risk of Experiencing a Resuscitated Cardiac Arrest Included in the POE
Description: For each subject, the time to first occurrence of a resuscitated cardiac arrest included in the POE was evaluated using time-to-event analysis.
Time Frame: From randomization up to 6 years
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Randomized Sibutramine | Randomized Placebo
Number analyzed (Participants) | 4906 | 4898
Participants | 11 | 7
Statistical Analysis 1: Comparison: Randomized Sibutramine vs Randomized Placebo; Test type: Superiority or Other; p = 0.343, Log Rank; Cox Proportional Hazard = 1.582, 95% CI 2-sided [0.613 to 4.081]

7. Secondary Outcome: Risk of Experiencing Cardiovascular Death Included in the POE
Description: For each subject, the time to cardiovascular death included in the POE was evaluated using time-to-event analysis.
Time Frame: From randomization up to 6 years
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Randomized Sibutramine | Randomized Placebo
Number analyzed (Participants) | 4906 | 4898
Participants | 223 | 229
Statistical Analysis 1: Comparison: Randomized Sibutramine vs Randomized Placebo; Test type: Superiority or Other; p = 0.899, Log Rank; Cox Proportional Hazard = 0.988, 95% CI 2-sided [0.822 to 1.188]

ADVERSE EVENTS:
Time Frame: Treatment-emergent serious adverse events (SAE) were defined as those that began on or after the first dose of randomized study drug (sibutramine or placebo) during the Randomization Phase through 30 days after the last dose.
Description: SAEs confirmed to be outcome events are included.
  Lead-in Period SAEs occurring on or after the first dose of sibutramine during the Lead-in Period through 30 days after the last dose of sibutramine for subjects who discontinued or through 30 days into the Randomization Phase for subjects who were randomized are included.
Groups:
- Lead-in Period Sibutramine: Subjects who received sibutramine 10 mg QD plus standard care for weight management during a 6-week Lead-in Period.
- Randomized Sibutramine: Subjects who successfully completed a 6-week Lead-in Period and who were randomized to receive sibutramine plus standard care for weight management during the Treatment Period of the Randomization Phase, and if sibutramine was prematurely discontinued, they received standard care for weight management during the Follow-up Period of the Randomization Phase.
- Randomized Placebo: Subjects who successfully completed a 6-week Lead-in Period and who were randomized to receive placebo plus standard care for weight management during the Treatment Period of the Randomizaiton Phase, and if placebo was prematurely discontinued, they received standard care for weight management during the Follow-up Period of the Randomization Phase.
Arm/Group | Lead-in Period Sibutramine | Randomized Sibutramine | Randomized Placebo
Serious Adverse Events (participants affected / at risk) | 425/10744 | 2063/4904 | 1977/4881
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lead-in Period Sibutramine (N=10744) | Randomized Sibutramine (N=4904) | Randomized Placebo (N=4881)
Anemia (Blood and lymphatic system disorders) | 0 | 19 | 11
Bicytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Coagulopathy (Blood and lymphatic system disorders) | 0 | 0 | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 0 | 1
Hemolytic anemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Hemorrhagic anemia (Blood and lymphatic system disorders) | 0 | 0 | 3
Hemorrhagic disorder (Blood and lymphatic system disorders) | 0 | 0 | 1
Hypersplenism (Blood and lymphatic system disorders) | 0 | 1 | 0
Hypochromic anemia (Blood and lymphatic system disorders) | 1 | 2 | 0
Hypoprothrombinanemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 1 | 0
Iron deficiency anemia (Blood and lymphatic system disorders) | 0 | 4 | 4
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 1 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0
Lymphatic obstruction (Blood and lymphatic system disorders) | 1 | 0 | 0
Lymphocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1
Microcytic anemia (Blood and lymphatic system disorders) | 0 | 2 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Normochromic normocytic anemia (Blood and lymphatic system disorders) | 0 | 2 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 6 | 25 | 26
Acute left ventricular failure (Cardiac disorders) | 0 | 3 | 3
Acute myocardial infarction (Cardiac disorders) | 3 | 87 | 87
Adams-Stokes syndrome (Cardiac disorders) | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 21 | 111 | 133
Angina unstable (Cardiac disorders) | 23 | 122 | 104
Aortic valve disease (Cardiac disorders) | 1 | 2 | 0
Aortic valve disease mixed (Cardiac disorders) | 0 | 4 | 2
Aortic valve incompetence (Cardiac disorders) | 0 | 3 | 1
Aortic valve stenosis (Cardiac disorders) | 0 | 7 | 9
Arrhythmia (Cardiac disorders) | 0 | 0 | 6
Arrhythmia supraventricular (Cardiac disorders) | 0 | 1 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 4 | 8
Atrial fibrillation (Cardiac disorders) | 20 | 115 | 135
Atrial flutter (Cardiac disorders) | 4 | 21 | 29
Atrial tachycardia (Cardiac disorders) | 0 | 1 | 0
Atrial thrombosis (Cardiac disorders) | 0 | 2 | 0
Atrioventricular block (Cardiac disorders) | 1 | 2 | 1
Atrioventricular block complete (Cardiac disorders) | 2 | 8 | 16
Atrioventricular block first degree (Cardiac disorders) | 0 | 1 | 2
Atrioventricular block second degree (Cardiac disorders) | 0 | 3 | 16
Bradyarrhythmia (Cardiac disorders) | 0 | 2 | 3
Bradycardia (Cardiac disorders) | 1 | 7 | 7
Bundle branch block right (Cardiac disorders) | 0 | 1 | 1
Cardiac aneurysm (Cardiac disorders) | 0 | 2 | 0
Cardiac arrest (Cardiac disorders) | 0 | 24 | 14
Cardiac asthma (Cardiac disorders) | 0 | 1 | 1
Cardiac disorder (Cardiac disorders) | 0 | 1 | 1
Cardiac failure (Cardiac disorders) | 2 | 82 | 80
Cardiac failure acute (Cardiac disorders) | 0 | 3 | 9
Cardiac failure chronic (Cardiac disorders) | 0 | 5 | 8
Cardiac failure congestive (Cardiac disorders) | 3 | 53 | 41
Cardiac tamponade (Cardiac disorders) | 0 | 2 | 1
Cardio-respiratory arrest (Cardiac disorders) | 1 | 1 | 2
Cardiogenic shock (Cardiac disorders) | 0 | 4 | 5
Cardiomyopathy (Cardiac disorders) | 0 | 1 | 1
Cardiopulmonary failure (Cardiac disorders) | 0 | 3 | 2
Cardiovascular insufficiency (Cardiac disorders) | 0 | 1 | 0
Chronic right ventricular failure (Cardiac disorders) | 0 | 0 | 1
Conduction disorder (Cardiac disorders) | 0 | 1 | 1
Congestive cardiomyopathy (Cardiac disorders) | 1 | 7 | 6
Cor pulmonale chronic (Cardiac disorders) | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 15 | 135 | 118
Coronary artery dissection (Cardiac disorders) | 0 | 1 | 0
Coronary artery insufficiency (Cardiac disorders) | 0 | 3 | 3
Coronary artery occlusion (Cardiac disorders) | 1 | 3 | 8
Coronary artery stenosis (Cardiac disorders) | 4 | 76 | 74
Coronary artery thrombosis (Cardiac disorders) | 1 | 2 | 2
Diastolic dysfunction (Cardiac disorders) | 0 | 0 | 1
Extrasystoles (Cardiac disorders) | 0 | 0 | 1
Hypertensive cardiomyopathy (Cardiac disorders) | 0 | 0 | 1
Hypertensive heart disease (Cardiac disorders) | 0 | 1 | 1
Intracardiac thrombus (Cardiac disorders) | 0 | 1 | 2
Ischemic cardiomyopathy (Cardiac disorders) | 0 | 10 | 13
Left ventricular dysfunction (Cardiac disorders) | 0 | 1 | 3
Left ventricular failure (Cardiac disorders) | 1 | 10 | 16
Left ventricular hypertrophy (Cardiac disorders) | 1 | 0 | 0
Mitral valve incompetence (Cardiac disorders) | 0 | 4 | 6
Mitral valve stenosis (Cardiac disorders) | 0 | 1 | 1
Myocardial infarction (Cardiac disorders) | 11 | 87 | 80
Myocardial ischemia (Cardiac disorders) | 5 | 57 | 36
Nodal arrhythmia (Cardiac disorders) | 0 | 0 | 1
Palpitations (Cardiac disorders) | 3 | 2 | 6
Pericardial effusion (Cardiac disorders) | 0 | 0 | 2
Pericarditis (Cardiac disorders) | 0 | 2 | 1
Postinfarction angina (Cardiac disorders) | 0 | 0 | 1
Prinzmetal angina (Cardiac disorders) | 0 | 0 | 1
Right ventricular failure (Cardiac disorders) | 0 | 4 | 3
Sick sinus syndrome (Cardiac disorders) | 2 | 11 | 12
Silent myocardial infarction (Cardiac disorders) | 0 | 5 | 4
Sinoatrial block (Cardiac disorders) | 0 | 2 | 1
Sinus arrhythmia (Cardiac disorders) | 0 | 1 | 3
Sinus bradycardia (Cardiac disorders) | 0 | 2 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1
Subendocardial ischemia (Cardiac disorders) | 0 | 1 | 0
Supraventricular extrasystoles (Cardiac disorders) | 0 | 0 | 2
Supraventricular tachyarrhythmia (Cardiac disorders) | 0 | 3 | 0
Supraventricular tachycardia (Cardiac disorders) | 3 | 12 | 6
Tachyarrhythmia (Cardiac disorders) | 0 | 3 | 2
Tachycardia (Cardiac disorders) | 0 | 0 | 2
Torsade de pointes (Cardiac disorders) | 0 | 1 | 0
Tricuspid valve incompetence (Cardiac disorders) | 0 | 1 | 0
Trifascicular block (Cardiac disorders) | 2 | 0 | 0
Ventricular arrhythmia (Cardiac disorders) | 0 | 3 | 1
Ventricular extrasystoles (Cardiac disorders) | 0 | 7 | 2
Ventricular failure (Cardiac disorders) | 0 | 0 | 1
Ventricular fibrillation (Cardiac disorders) | 2 | 5 | 6
Ventricular tachyarrhythmia (Cardiac disorders) | 0 | 2 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 25 | 18
Atrial septal defect (Congenital, familial and genetic disorders) | 0 | 0 | 1
Congenital cystic kidney disease (Congenital, familial and genetic disorders) | 0 | 0 | 1
Congenital spondylolithesis (Congenital, familial and genetic disorders) | 1 | 0 | 0
Dysplastic naevus syndrome (Congenital, familial and genetic disorders) | 0 | 1 | 0
Gastrointestinal angiodysplasia (Congenital, familial and genetic disorders) | 0 | 1 | 0
Gastrointestinal angiodysplasia hemorrhagic (Congenital, familial and genetic disorders) | 0 | 0 | 1
Hydrocele (Congenital, familial and genetic disorders) | 2 | 1 | 0
Phimosis (Congenital, familial and genetic disorders) | 0 | 1 | 3
Acute vestibular syndrome (Ear and labyrinth disorders) | 0 | 2 | 0
Aural polyp (Ear and labyrinth disorders) | 0 | 0 | 1
Deafness unilateral (Ear and labyrinth disorders) | 0 | 1 | 1
Hearing impaired (Ear and labyrinth disorders) | 0 | 0 | 1
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 1
Neurosensory hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 1
Sudden hearing loss (Ear and labyrinth disorders) | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 4 | 5
Vertigo positional (Ear and labyrinth disorders) | 0 | 2 | 2
Vestibular disorder (Ear and labyrinth disorders) | 0 | 3 | 0
Autoimmune thyroiditis (Endocrine disorders) | 0 | 0 | 1
Goiter (Endocrine disorders) | 0 | 7 | 6
Hyperparathyroidism (Endocrine disorders) | 0 | 3 | 0
Hyperparathyroidism primary (Endocrine disorders) | 1 | 0 | 2
Hyperthyroidism (Endocrine disorders) | 0 | 5 | 5
Hypothyroidism (Endocrine disorders) | 0 | 0 | 1
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 1 | 0
Myxedema (Endocrine disorders) | 0 | 0 | 1
Toxic nodular goiter (Endocrine disorders) | 1 | 1 | 1
Amaurosis (Eye disorders) | 0 | 1 | 0
Angle closure glaucoma (Eye disorders) | 0 | 1 | 2
Aphakia (Eye disorders) | 0 | 0 | 1
Cataract (Eye disorders) | 4 | 33 | 29
Cataract diabetic (Eye disorders) | 0 | 0 | 1
Cataract nuclear (Eye disorders) | 1 | 0 | 2
Cataract subcapsular (Eye disorders) | 0 | 2 | 0
Diabetic retinopathy (Eye disorders) | 0 | 6 | 4
Diplopia (Eye disorders) | 1 | 1 | 0
Extraocular muscle paresis (Eye disorders) | 1 | 0 | 0
Eye hemorrhage (Eye disorders) | 0 | 1 | 1
Eye pain (Eye disorders) | 1 | 0 | 0
Glaucoma (Eye disorders) | 0 | 1 | 3
Iris bombe (Eye disorders) | 0 | 0 | 1
Keratitis (Eye disorders) | 0 | 1 | 0
Lens dislocation (Eye disorders) | 0 | 0 | 1
Macular hole (Eye disorders) | 0 | 1 | 0
Macular edema (Eye disorders) | 0 | 1 | 0
Maculopathy (Eye disorders) | 0 | 1 | 0
Ocular myasthenia (Eye disorders) | 0 | 1 | 0
Ocular vascular disorder (Eye disorders) | 0 | 0 | 1
Open-angle glaucoma (Eye disorders) | 0 | 2 | 1
Optic ischemic neuropathy (Eye disorders) | 1 | 1 | 0
Punctate keratitis (Eye disorders) | 1 | 0 | 0
Retinal artery occlusion (Eye disorders) | 0 | 1 | 3
Retinal detachment (Eye disorders) | 0 | 10 | 5
Retinal hemorrhage (Eye disorders) | 1 | 2 | 0
Retinal vein occlusion (Eye disorders) | 0 | 0 | 1
Retinal vein thrombosis (Eye disorders) | 0 | 1 | 0
Strabismus (Eye disorders) | 0 | 1 | 0
Synchysis scintillans (Eye disorders) | 0 | 0 | 1
Ulcerative keratitis (Eye disorders) | 0 | 1 | 0
Uveitis (Eye disorders) | 0 | 1 | 0
Visual impairment (Eye disorders) | 0 | 0 | 1
Vitreous detachment (Eye disorders) | 0 | 1 | 0
Vitreous disorder (Eye disorders) | 1 | 0 | 0
Vitreous hemorrhage (Eye disorders) | 0 | 0 | 3
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 0 | 7 | 3
Abdominal hernia obstructive (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal mass (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 8 | 9
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2 | 6
Abdominal strangulated hernia (Gastrointestinal disorders) | 0 | 0 | 2
Anal fissure (Gastrointestinal disorders) | 0 | 3 | 2
Anal fistula (Gastrointestinal disorders) | 0 | 3 | 2
Anal stenosis (Gastrointestinal disorders) | 0 | 1 | 1
Anal ulcer (Gastrointestinal disorders) | 0 | 0 | 1
Barrett's esophagus (Gastrointestinal disorders) | 0 | 1 | 1
Cecitis (Gastrointestinal disorders) | 0 | 0 | 1
Change of bowel habit (Gastrointestinal disorders) | 0 | 1 | 0
Celiac artery stenosis (Gastrointestinal disorders) | 0 | 0 | 2
Colitis (Gastrointestinal disorders) | 0 | 5 | 0
Colitis ischemic (Gastrointestinal disorders) | 0 | 2 | 2
Colonic polyp (Gastrointestinal disorders) | 2 | 3 | 10
Constipation (Gastrointestinal disorders) | 1 | 5 | 4
Diabetic gastroparesis (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 4 | 7
Diarrhea hemorrhagic (Gastrointestinal disorders) | 1 | 0 | 0
Diverticulitis intestinal hemorrhagic (Gastrointestinal disorders) | 1 | 1 | 0
Diverticulum (Gastrointestinal disorders) | 1 | 2 | 2
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 2 | 5
Diverticulum intestinal hemorrhagic (Gastrointestinal disorders) | 0 | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 5 | 4
Duodenal ulcer hemorrhage (Gastrointestinal disorders) | 0 | 12 | 2
Duodenal ulcer perforation (Gastrointestinal disorders) | 0 | 1 | 0
Duodenitis (Gastrointestinal disorders) | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 4 | 3
Enteritis (Gastrointestinal disorders) | 0 | 0 | 3
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 1
Erosive esophagitis (Gastrointestinal disorders) | 0 | 1 | 0
Fecal incontinence (Gastrointestinal disorders) | 0 | 0 | 1
Fecaloma (Gastrointestinal disorders) | 1 | 3 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 1 | 1
Gastric hemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Gastric mucosal lesion (Gastrointestinal disorders) | 0 | 0 | 1
Gastric perforation (Gastrointestinal disorders) | 0 | 0 | 1
Gastric polyps (Gastrointestinal disorders) | 0 | 4 | 2
Gastric ulcer (Gastrointestinal disorders) | 3 | 5 | 7
Gastric ulcer hemorrhage (Gastrointestinal disorders) | 0 | 9 | 9
Gastritis (Gastrointestinal disorders) | 0 | 8 | 4
Gastritis atrophic (Gastrointestinal disorders) | 0 | 1 | 0
Gastritis erosive (Gastrointestinal disorders) | 0 | 4 | 3
Gastritis hemorrhagic (Gastrointestinal disorders) | 1 | 2 | 5
Gastroduodenitis (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 3 | 4
Gastrointestinal inflammation (Gastrointestinal disorders) | 2 | 1 | 1
Gastrointestinal ulcer hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 4 | 6
Gastroesophageal sphincter insufficiency (Gastrointestinal disorders) | 0 | 0 | 1
Gastroesophagitis (Gastrointestinal disorders) | 1 | 1 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 1
Hematochezia (Gastrointestinal disorders) | 0 | 1 | 0
Hemorrhagic erosive gastritis (Gastrointestinal disorders) | 0 | 1 | 0
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Hemorrhoids (Gastrointestinal disorders) | 1 | 3 | 4
Hernial eventration (Gastrointestinal disorders) | 0 | 5 | 2
Hiatus hernia (Gastrointestinal disorders) | 0 | 3 | 2
Ileitis (Gastrointestinal disorders) | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 4 | 2
Ileus paralytic (Gastrointestinal disorders) | 0 | 1 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 4 | 13 | 18
Intestinal ischemia (Gastrointestinal disorders) | 0 | 4 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 6 | 3
Intra-abdominal hematoma (Gastrointestinal disorders) | 0 | 1 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 1 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 0 | 1
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 2
Mechanical ileus (Gastrointestinal disorders) | 0 | 1 | 1
Melena (Gastrointestinal disorders) | 1 | 0 | 1
Melanosis coli (Gastrointestinal disorders) | 0 | 0 | 1
Mesenteric artery stenosis (Gastrointestinal disorders) | 0 | 0 | 2
Mesenteric artery thrombosis (Gastrointestinal disorders) | 0 | 0 | 1
Mesenteric occlusion (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 2 | 5
Esophageal stenosis (Gastrointestinal disorders) | 0 | 0 | 1
Esophageal ulcer hemorrhage (Gastrointestinal disorders) | 0 | 1 | 1
Esophagitis (Gastrointestinal disorders) | 3 | 5 | 1
Esophagitis ulcerative (Gastrointestinal disorders) | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 3 | 4
Pancreatitis acute (Gastrointestinal disorders) | 0 | 3 | 14
Pancreatitis chronic (Gastrointestinal disorders) | 0 | 1 | 1
Pancreatitis necrotizing (Gastrointestinal disorders) | 0 | 0 | 1
Papilla of Vater stenosis (Gastrointestinal disorders) | 0 | 0 | 1
Peptic ulcer (Gastrointestinal disorders) | 0 | 2 | 3
Peptic ulcer hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Periodontal disease (Gastrointestinal disorders) | 0 | 1 | 0
Peritoneal adhesions (Gastrointestinal disorders) | 0 | 0 | 1
Peritoneal hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Peritonitis (Gastrointestinal disorders) | 0 | 1 | 2
Proctitis (Gastrointestinal disorders) | 0 | 0 | 1
Rectal hemorrhage (Gastrointestinal disorders) | 1 | 2 | 2
Rectal perforation (Gastrointestinal disorders) | 0 | 0 | 1
Rectal polyp (Gastrointestinal disorders) | 0 | 2 | 2
Rectal prolapse (Gastrointestinal disorders) | 0 | 1 | 0
Reflux esophagitis (Gastrointestinal disorders) | 0 | 0 | 1
Retroperitoneal fibrosis (Gastrointestinal disorders) | 0 | 1 | 0
Retroperitoneal hematoma (Gastrointestinal disorders) | 0 | 1 | 1
Small intestinal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Subileus (Gastrointestinal disorders) | 0 | 1 | 0
Tongue hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Tooth disorder (Gastrointestinal disorders) | 0 | 0 | 1
Tooth loss (Gastrointestinal disorders) | 0 | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 12 | 9
Umbilical hernia, obstructive (Gastrointestinal disorders) | 0 | 0 | 1
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 3 | 3
Varices esophageal (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 5
Abasia (General disorders) | 0 | 1 | 0
Adhesion (General disorders) | 0 | 1 | 0
Adverse drug reaction (General disorders) | 0 | 1 | 2
Asthenia (General disorders) | 0 | 3 | 1
Catheter-related complication (General disorders) | 0 | 0 | 1
Chest discomfort (General disorders) | 1 | 2 | 2
Chest pain (General disorders) | 5 | 22 | 18
Chills (General disorders) | 0 | 0 | 2
Cyst (General disorders) | 0 | 1 | 0
Death (General disorders) | 17 | 25 | 18
Drug intolerance (General disorders) | 0 | 0 | 1
Dysplasia (General disorders) | 0 | 0 | 2
Fatigue (General disorders) | 1 | 2 | 5
Foaming at mouth (General disorders) | 0 | 0 | 1
General physical health deterioration (General disorders) | 0 | 1 | 0
Hernia obstructive (General disorders) | 1 | 1 | 1
Impaired healing (General disorders) | 0 | 1 | 0
Implant expulsion (General disorders) | 0 | 0 | 1
Implant site fibrosis (General disorders) | 0 | 1 | 0
Implant site inflammation (General disorders) | 0 | 0 | 1
Inflammation (General disorders) | 0 | 0 | 2
Malaise (General disorders) | 0 | 2 | 3
Mechanical complication of implant (General disorders) | 0 | 2 | 0
Metaplasia (General disorders) | 0 | 0 | 1
Multi-organ failure (General disorders) | 1 | 3 | 2
Necrosis (General disorders) | 0 | 0 | 2
Non-cardiac chest pain (General disorders) | 2 | 19 | 15
Pain (General disorders) | 2 | 2 | 0
Peripheral edema (General disorders) | 0 | 4 | 3
Pyrexia (General disorders) | 0 | 5 | 5
Sudden cardiac death (General disorders) | 0 | 11 | 4
Sudden death (General disorders) | 3 | 19 | 26
Swelling (General disorders) | 0 | 0 | 1
Autoimmune hepatitis (Hepatobiliary disorders) | 0 | 0 | 1
Bile duct obstruction (Hepatobiliary disorders) | 0 | 0 | 1
Bile duct stenosis (Hepatobiliary disorders) | 0 | 0 | 1
Bile duct stone (General disorders) | 0 | 0 | 1
Biliary cirrhosis primary (Hepatobiliary disorders) | 0 | 1 | 1
Biliary colic (Hepatobiliary disorders) | 1 | 1 | 2
Cholangitis (Hepatobiliary disorders) | 0 | 1 | 4
Cholangitis acute (Hepatobiliary disorders) | 0 | 1 | 1
Cholecystitis (Hepatobiliary disorders) | 2 | 8 | 7
Cholecystitis acute (Hepatobiliary disorders) | 0 | 7 | 5
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 1 | 4
Cholelithiasis (Hepatobiliary disorders) | 2 | 26 | 25
Cirrhosis alcoholic (Hepatobiliary disorders) | 1 | 0 | 1
Gallbladder cholesterolosis (Hepatobiliary disorders) | 0 | 0 | 1
Gallbladder disorder (Hepatobiliary disorders) | 1 | 0 | 1
Gallbladder obstruction (Hepatobiliary disorders) | 0 | 0 | 1
Gallbladder perforation (Hepatobiliary disorders) | 0 | 0 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 2 | 0
Hepatic lesion (General disorders) | 0 | 1 | 0
Hepatic mass (Hepatobiliary disorders) | 0 | 1 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 1
Hepatitis acute (Hepatobiliary disorders) | 0 | 1 | 0
Hepatorenal failure (Hepatobiliary disorders) | 0 | 0 | 1
Liver disorder (Hepatobiliary disorders) | 1 | 1 | 0
Liver injury (Hepatobiliary disorders) | 0 | 0 | 1
Anaphylactic reaction (Immune system disorders) | 0 | 1 | 1
Anaphylactic shock (Immune system disorders) | 1 | 4 | 1
Hypersensitivity (Immune system disorders) | 0 | 4 | 3
Abdominal abscess (Infections and infestations) | 0 | 0 | 1
Abscess limb (Infections and infestations) | 0 | 2 | 2
Abscess neck (Infections and infestations) | 0 | 1 | 0
Abscess oral (Infections and infestations) | 0 | 0 | 1
Acarodermatitis (Infections and infestations) | 0 | 0 | 1
Anal abscess (Infections and infestations) | 1 | 1 | 3
Appendicitis (Infections and infestations) | 0 | 6 | 3
Appendicitis perforated (Infections and infestations) | 0 | 1 | 0
Arteriosclerotic gangrene (Infections and infestations) | 0 | 0 | 2
Arthritis bacterial (Infections and infestations) | 0 | 1 | 1
Arthritis infective (Infections and infestations) | 0 | 1 | 0
Bacterial infection (Infections and infestations) | 0 | 1 | 0
Bacterial pyelonephritis (Infections and infestations) | 0 | 1 | 0
Biliary sepsis (Infections and infestations) | 0 | 1 | 1
Bronchiectasis (Infections and infestations) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 13 | 15
Bronchitis bacterial (Infections and infestations) | 0 | 1 | 0
Bronchitis viral (Infections and infestations) | 0 | 1 | 1
Bronchopneumonia (Infections and infestations) | 2 | 14 | 17
Bronchopulmonary aspergillosis allergic (Infections and infestations) | 0 | 1 | 0
Campylobacter intestinal infection (Infections and infestations) | 0 | 2 | 0
Catheter-site infection (Infections and infestations) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 3 | 19 | 17
Cellulitis staphylococcal (Infections and infestations) | 0 | 0 | 1
Central line infection (Infections and infestations) | 0 | 0 | 1
Cholecystitis infective (Infections and infestations) | 0 | 3 | 4
Chronic sinusitis (Infections and infestations) | 0 | 2 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 1 | 0
Cystitis (Infections and infestations) | 1 | 7 | 2
Dengue fever (Infections and infestations) | 0 | 0 | 1
Device-related infection (Infections and infestations) | 0 | 2 | 3
Diabetic foot infection (Infections and infestations) | 0 | 7 | 6
Diabetic gangrene (Infections and infestations) | 2 | 8 | 4
Diarrhea infectious (Infections and infestations) | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 7 | 8
Endocarditis (Infections and infestations) | 0 | 2 | 4
Endocarditis bacterial (Infections and infestations) | 0 | 2 | 0
Endocarditis staphylococcal (Infections and infestations) | 0 | 1 | 0
Endophthalmitis (Infections and infestations) | 0 | 1 | 0
Entereocolitis viral (Infections and infestations) | 0 | 1 | 0
Erysipelas (Infections and infestations) | 5 | 23 | 14
Escherichia sepsis (Infections and infestations) | 0 | 3 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 1
Eye infection (Infections and infestations) | 0 | 1 | 0
Furuncle (Infections and infestations) | 0 | 2 | 0
Gallbladder empyema (Infections and infestations) | 0 | 0 | 1
Gangrene (Infections and infestations) | 3 | 3 | 5
Gastroenteritis (Infections and infestations) | 4 | 13 | 15
Gastroenteritis bacterial (Infections and infestations) | 1 | 1 | 0
Gastroenteritis clostridial (Infections and infestations) | 0 | 0 | 2
Gastroenteritis rotavirus (Infections and infestations) | 0 | 2 | 0
Gastroenteritis salmonella (Infections and infestations) | 0 | 1 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 2 | 3
Gingival abscess (Infections and infestations) | 0 | 0 | 1
Graft infection (Infections and infestations) | 0 | 0 | 1
Groin abscess (Infections and infestations) | 1 | 1 | 2
Hematoma infection (Infections and infestations) | 0 | 1 | 0
Helicobacter infection (Infections and infestations) | 0 | 0 | 1
Hepatitis A (Infections and infestations) | 0 | 1 | 0
Hepatitis B (Infections and infestations) | 1 | 1 | 2
Hepatitis C (Infections and infestations) | 0 | 1 | 1
Hepatitis viral (Infections and infestations) | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 2 | 3 | 2
Herpes zoster ophthalmic (Infections and infestations) | 0 | 2 | 1
Infected sebaceous cyst (Infections and infestations) | 0 | 0 | 1
Infected skin ulcer (Infections and infestations) | 1 | 7 | 2
Infection (Infections and infestations) | 0 | 0 | 3
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 | 7 | 12
Infective tenosynovitis (Infections and infestations) | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 1 | 0
Infusion site infection (Infections and infestations) | 1 | 1 | 0
Intervertebral discitis (Infections and infestations) | 0 | 0 | 1
Kidney infection (Infections and infestations) | 0 | 0 | 1
Klebsiella sepsis (Infections and infestations) | 0 | 0 | 1
Labyrinthitis (Infections and infestations) | 0 | 1 | 1
Laryngitis (Infections and infestations) | 0 | 0 | 1
Liver abscess (Infections and infestations) | 0 | 0 | 1
Lobar pneumonia (Infections and infestations) | 0 | 13 | 6
Localized infection (Infections and infestations) | 0 | 3 | 4
Lower respiratory tract infection (Infections and infestations) | 1 | 4 | 10
Lung abscess (Infections and infestations) | 0 | 1 | 1
Lung infection (Infections and infestations) | 0 | 3 | 3
Lung infection pseudomonal (Infections and infestations) | 0 | 0 | 1
Lyme disease (Infections and infestations) | 0 | 3 | 1
Lymph node tuberculosis (Infections and infestations) | 0 | 1 | 0
Mastitis (Infections and infestations) | 0 | 0 | 1
Mediastinitis (Infections and infestations) | 0 | 4 | 1
Meningococcal sepsis (Infections and infestations) | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1
Neuroborreliosis (Infections and infestations) | 1 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 1 | 0
Orchitis (Infections and infestations) | 1 | 2 | 0
Osteomyelitis (Infections and infestations) | 3 | 13 | 4
Otitis media acute (Infections and infestations) | 0 | 2 | 1
Otitis media chronic (Infections and infestations) | 1 | 0 | 0
Paronychia (Infections and infestations) | 0 | 1 | 0
Parotitis (Infections and infestations) | 0 | 1 | 1
Perihepatic abscess (Infections and infestations) | 0 | 0 | 1
Perineal abscess (Infections and infestations) | 0 | 0 | 2
Perirectal abscess (Infections and infestations) | 0 | 1 | 0
Peritonsillar abscess (Infections and infestations) | 0 | 1 | 1
Peritonsillitis (Infections and infestations) | 0 | 1 | 0
Pharyngeal abscess (Infections and infestations) | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 0
Pleurisy viral (Infections and infestations) | 1 | 0 | 0
Pneumococcal sepsis (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 5 | 51 | 59
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 3
Pneumonia escherichia (Infections and infestations) | 0 | 1 | 1
Pneumonia legionella (Infections and infestations) | 0 | 0 | 2
Pneumonia pneumococcal (Infections and infestations) | 0 | 0 | 1
Post-procedural cellulitis (Infections and infestations) | 0 | 1 | 0
Post-procedural infection (Infections and infestations) | 1 | 4 | 2
Postoperative abscess (Infections and infestations) | 0 | 1 | 1
Postoperative wound infection (Infections and infestations) | 0 | 3 | 6
Prostatic abscess (Infections and infestations) | 0 | 1 | 0
Pulmonary sepsis (Infections and infestations) | 0 | 1 | 0
Pulmonary tuberculosis (Infections and infestations) | 0 | 1 | 2
Pyelocystitis (Infections and infestations) | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 6 | 8
Pyelonephritis acute (Infections and infestations) | 1 | 1 | 3
Pyothorax (Infections and infestations) | 0 | 1 | 0
Rash pustular (Infections and infestations) | 0 | 1 | 0
Rectal abscess (Infections and infestations) | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 7 | 8
Salmonella sepsis (Infections and infestations) | 0 | 1 | 0
Salmonellosis (Infections and infestations) | 3 | 0 | 1
Sepsis (Infections and infestations) | 0 | 11 | 13
Septic shock (Infections and infestations) | 0 | 9 | 6
Sinusitis (Infections and infestations) | 0 | 2 | 0
Sinusitis bacterial (Infections and infestations) | 0 | 1 | 0
Skin bacterial infection (Infections and infestations) | 0 | 1 | 0
Skin infection (Infections and infestations) | 0 | 2 | 0
Staphylococcal infection (Infections and infestations) | 1 | 3 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 3 | 2
Sternitis (Infections and infestations) | 0 | 1 | 0
Streptococcal sepsis (Infections and infestations) | 0 | 1 | 0
Subacute endocarditis (Infections and infestations) | 0 | 1 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 2 | 1
Sweat gland infection (Infections and infestations) | 1 | 0 | 1
Testicular abscess (Infections and infestations) | 0 | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 0 | 1
Toxic shock syndrome (Infections and infestations) | 1 | 0 | 0
Tracheitis (Infections and infestations) | 0 | 2 | 0
Tracheobronchitis (Infections and infestations) | 0 | 0 | 2
Tuberculosis (Infections and infestations) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 4 | 1
Urinary tract infection (Infections and infestations) | 0 | 16 | 23
Urinary tract infection bacterial (Infections and infestations) | 0 | 0 | 1
Urosepsis (Infections and infestations) | 0 | 6 | 3
Vestibular neuronitis (Infections and infestations) | 0 | 2 | 2
Viral infection (Infections and infestations) | 0 | 1 | 3
Viral labyrinthitis (Infections and infestations) | 0 | 0 | 2
Visceral leishmaniasis (Infections and infestations) | 0 | 0 | 1
Vulval cellulitis (Infections and infestations) | 0 | 1 | 0
Wound abscess (Infections and infestations) | 0 | 1 | 0
Wound infection (Infections and infestations) | 0 | 2 | 3
Wound infection staphylococcal (Infections and infestations) | 0 | 4 | 1
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1 | 0
Accidental needle stick (Injury, poisoning and procedural complications) | 0 | 0 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 2 | 1
Anastomotic complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 4 | 4
Arterial restenosis (Injury, poisoning and procedural complications) | 0 | 2 | 1
Ateriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 0 | 1 | 0
Asbestosis (Injury, poisoning and procedural complications) | 0 | 0 | 1
Bladder injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Brachial plexus injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Brain contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Cardiac pacemaker malfunction (Injury, poisoning and procedural complications) | 0 | 3 | 3
Cerebral hemorrhage traumatic (Injury, poisoning and procedural complications) | 1 | 1 | 0
Cerebral hyperperfusion syndrome (Injury, poisoning and procedural complications) | 0 | 0 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 3 | 1
Confusion postoperative (Injury, poisoning and procedural complications) | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 3 | 3
Coronary artery restenosis (Injury, poisoning and procedural complications) | 3 | 10 | 11
Coronary bypass thrombosis (Injury, poisoning and procedural complications) | 0 | 1 | 0
Device breakage (Injury, poisoning and procedural complications) | 0 | 0 | 2
Device dislocation (Injury, poisoning and procedural complications) | 0 | 1 | 0
Device failure (Injury, poisoning and procedural complications) | 1 | 5 | 5
Device lead damage (Injury, poisoning and procedural complications) | 0 | 0 | 1
Device malfunction (Injury, poisoning and procedural complications) | 0 | 1 | 2
Device occlusion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Dislocation of joint prosthesis (Injury, poisoning and procedural complications) | 0 | 2 | 2
Drug administration error (Injury, poisoning and procedural complications) | 0 | 0 | 1
Drug dispensing error (Injury, poisoning and procedural complications) | 0 | 1 | 0
Drug toxicity (Injury, poisoning and procedural complications) | 0 | 0 | 1
Eye injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Face injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 4 | 5
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 2 | 5
Femur fracture (Injury, poisoning and procedural complications) | 0 | 3 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 1 | 4
Forearm fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0
Foreign body trauma (Injury, poisoning and procedural complications) | 0 | 1 | 1
Fracture displacement (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fractured sacrum (Injury, poisoning and procedural complications) | 0 | 1 | 0
Gastroenteritis radiation (Injury, poisoning and procedural complications) | 0 | 2 | 1
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0 | 0 | 1
Graft thrombosis (Injury, poisoning and procedural complications) | 0 | 5 | 2
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 1 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 6
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 4
Iatrogenic injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Implantable defibrillator malfunction (Injury, poisoning and procedural complications) | 0 | 1 | 0
In-stent arterial restenosis (Injury, poisoning and procedural complications) | 0 | 2 | 5
In-stent coronary artery restenosis (Injury, poisoning and procedural complications) | 0 | 8 | 6
Inappropriate device stimulation of tissue (Injury, poisoning and procedural complications) | 0 | 0 | 1
Incision site complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 3 | 6
Incisional hernia, obstructive (Injury, poisoning and procedural complications) | 0 | 1 | 0
Injury (Injury, poisoning and procedural complications) | 1 | 6 | 4
Intervertebral disc injury (Injury, poisoning and procedural complications) | 0 | 0 | 2
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 3 | 8
Joint injury (Injury, poisoning and procedural complications) | 0 | 2 | 2
Joint sprain (Injury, poisoning and procedural complications) | 0 | 1 | 1
Keratorhexis (Injury, poisoning and procedural complications) | 0 | 1 | 0
Lead dislodgement (Injury, poisoning and procedural complications) | 0 | 0 | 1
Ligament rupture (Injury, poisoning and procedural complications) | 1 | 4 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Limb traumatic amputation (Injury, poisoning and procedural complications) | 0 | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 2 | 2
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 2 | 3
Medical device complication (Injury, poisoning and procedural complications) | 0 | 2 | 4
Medical device pain (Injury, poisoning and procedural complications) | 0 | 3 | 0
Meniscus lesion (Injury, poisoning and procedural complications) | 4 | 5 | 6
Multiple fractures (Injury, poisoning and procedural complications) | 0 | 0 | 1
Multiple injuries (Injury, poisoning and procedural complications) | 1 | 2 | 6
Muscle injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Muscle rupture (Injury, poisoning and procedural complications) | 0 | 2 | 0
Operative hemorrhage (Injury, poisoning and procedural complications) | 0 | 2 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 2 | 0
Patella fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 1 | 1
Periprosthetic osteolysis (Injury, poisoning and procedural complications) | 0 | 1 | 0
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 0 | 1 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 4 | 4
Post procedural fistula (Injury, poisoning and procedural complications) | 0 | 0 | 1
Post procedural hematoma (Injury, poisoning and procedural complications) | 0 | 4 | 4
Post procedural hemorrhage (Injury, poisoning and procedural complications) | 2 | 5 | 2
Post procedural myocardial infarction (Injury, poisoning and procedural complications) | 0 | 1 | 0
Post procedural stroke (Injury, poisoning and procedural complications) | 0 | 1 | 0
Post procedural swelling (Injury, poisoning and procedural complications) | 0 | 0 | 1
Postmastectomy lymphedema syndrome (Injury, poisoning and procedural complications) | 0 | 1 | 0
Postoperative adhesion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Postoperative hernia (Injury, poisoning and procedural complications) | 0 | 0 | 1
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 2 | 3 | 3
Postoperative thrombosis (Injury, poisoning and procedural complications) | 0 | 1 | 0
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 | 1 | 0
Postpericardiotomy syndrome (Injury, poisoning and procedural complications) | 0 | 0 | 2
Procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 2
Procedural hypotension (Injury, poisoning and procedural complications) | 0 | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 3
Rib fracture (Injury, poisoning and procedural complications) | 0 | 2 | 3
Seroma (Injury, poisoning and procedural complications) | 0 | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 2 | 2
Skull fractured base (Injury, poisoning and procedural complications) | 0 | 1 | 0
Soft tissue injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 3 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Stent occlusion (Injury, poisoning and procedural complications) | 0 | 3 | 3
Sternal fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0
Subcutaneous hematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Subdural hematoma (Injury, poisoning and procedural complications) | 0 | 4 | 3
Tendon injury (Injury, poisoning and procedural complications) | 0 | 1 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 2 | 10
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 0 | 1 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Thrombosis in device (Injury, poisoning and procedural complications) | 0 | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1 | 2
Tongue injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Traumatic amputation (Injury, poisoning and procedural complications) | 0 | 1 | 0
Traumatic brain injury (Injury, poisoning and procedural complications) | 0 | 5 | 2
Traumatic fracture (Injury, poisoning and procedural complications) | 4 | 13 | 18
Traumatic hematoma (Injury, poisoning and procedural complications) | 0 | 3 | 1
Traumatic lung injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Traumatic shock (Injury, poisoning and procedural complications) | 0 | 1 | 0
Traumatic ulcer (Injury, poisoning and procedural complications) | 1 | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 3
Ureteric anastomosis complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Urinary retention postoperative (Injury, poisoning and procedural complications) | 0 | 1 | 1
Vaccination complication (Injury, poisoning and procedural complications) | 0 | 0 | 1
Vascular graft complication (Injury, poisoning and procedural complications) | 1 | 6 | 5
Vascular graft occlusion (Injury, poisoning and procedural complications) | 1 | 5 | 3
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 | 3 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1 | 1
Wound evisceration (Injury, poisoning and procedural complications) | 0 | 1 | 0
Wound hemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1
Wound necrosis (Injury, poisoning and procedural complications) | 0 | 3 | 2
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Angiogram (Investigations) | 0 | 0 | 2
Anticoagulation drug level above therapeutic (Investigations) | 0 | 1 | 1
Arteriogram coronary (Investigations) | 0 | 2 | 1
Arteriogram renal (Investigations) | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 1 | 0
Blood glucose increased (Investigations) | 0 | 1 | 1
Blood iron decreased (Investigations) | 0 | 0 | 1
Blood potassium decreased (Investigations) | 0 | 1 | 1
Body temperature increased (Investigations) | 1 | 0 | 0
Cardiac stress test abnormal (Investigations) | 0 | 2 | 1
Catheterization cardiac (Investigations) | 0 | 3 | 0
Coagulation time prolonged (Investigations) | 0 | 1 | 5
Colonoscopy (Investigations) | 0 | 1 | 1
Diagnostic procedure (Investigations) | 0 | 1 | 0
Ejection fraction decreased (Investigations) | 0 | 1 | 1
Hemoglobin decreased (Investigations) | 0 | 0 | 1
Heart rate irregular (Investigations) | 0 | 1 | 0
Hepatic enzyme increased (Investigations) | 0 | 1 | 0
International normalized ratio increased (Investigations) | 0 | 0 | 1
Investigation (Investigations) | 0 | 2 | 1
Laboratory test abnormal (Investigations) | 0 | 1 | 0
Medical observation (Investigations) | 0 | 0 | 1
Platelet count decreased (Investigations) | 0 | 1 | 0
Renal function test abnormal (Investigations) | 0 | 0 | 1
Scan myocardial perfusion abnormal (Investigations) | 0 | 1 | 1
Urine output decreased (Investigations) | 0 | 1 | 0
Weight decreased (Investigations) | 0 | 1 | 1
Weight increased (Investigations) | 0 | 4 | 2
X-ray abnormal (Investigations) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 5 | 5
Diabetes mellitus (Metabolism and nutrition disorders) | 3 | 30 | 28
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 4 | 67 | 50
Diabetes with hyperosmolarity (Metabolism and nutrition disorders) | 0 | 0 | 1
Diabetic foot (Metabolism and nutrition disorders) | 3 | 17 | 15
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 1
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 | 1 | 0
Gout (Metabolism and nutrition disorders) | 0 | 3 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 6 | 13
Hyperkalemia (Metabolism and nutrition disorders) | 3 | 6 | 5
Hyperphagia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 17 | 15
Hypokalemia (Metabolism and nutrition disorders) | 1 | 2 | 1
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypovolemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Insulin-requiring type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 2
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1 | 1
Metabolic disorder (Metabolism and nutrition disorders) | 0 | 2 | 0
Neuroglycopenia (Metabolism and nutrition disorders) | 0 | 1 | 0
Obesity (Metabolism and nutrition disorders) | 0 | 4 | 5
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 4 | 2
Weight loss poor (Metabolism and nutrition disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 7 | 10
Arthrofibrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 3 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 9 | 13
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Bunion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 4 | 3
Cervical spinal stenosis (Metabolism and nutrition disorders) | 0 | 0 | 1
Chondrocalcinosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Chrondopathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2
Exostosis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Facet joint syndrome (Metabolism and nutrition disorders) | 0 | 1 | 0
Fibromyalgia (Metabolism and nutrition disorders) | 1 | 0 | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 5 | 6
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Gouty tophus (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Hand deformity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 | 2 | 2
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 | 15 | 15
Intervertebral disc space narrowing (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Joint contracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Knee deformity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Ligament disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 9 | 12
Metatarsalgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Monarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscle hemorrhage (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 | 6 | 14
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 8 | 11
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 3 | 3
Myalgia intercostal (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 3 | 1
Osteitis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 9 | 107 | 88
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 4 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 6 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Patellofemoral pain syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 5 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 8 | 8
Scleroderma (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Senile ankylosing vertebral hyperostosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 6 | 6
Spinal disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 6 | 12
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2
Tendinous contracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Tendon calcification (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Acoustic neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Acute lymphocytic leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Acute myeloid leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 4
Anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Astrocytoma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 4
Basosquamous carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Benign anorectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Benign colonic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Benign lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 0
Benign neoplasm of bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3 | 1
Benign renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Benign salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 4
Bladder adenocarcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 7 | 6
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 2
Bladder cancer stage 0, with cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Bladder cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Bladder cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 2
Bladder papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 12 | 4
Bladder transitional cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 5 | 2
Bladder transitional cell carcinoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Bladder transitional cell carcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 20 | 15
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 5 | 2
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Breast cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Breast cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 2
Breast cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Breast cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Breast fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 4 | 0
Bronchioalveolar carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Chloroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 0
Chronic lymphocytic leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3 | 2
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 11 | 10
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 4 | 4
Colon cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Colon cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Colorectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 2
Endometrial cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Endometrial cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Follicle center lymphoma, follicular grade I, II, III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Gallbladder cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Gammopathy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 6 | 3
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Head and neck cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Intraductal papilloma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3 | 3
Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Leiomyosarcoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lentigo maligna stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Lip and/or oral cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Lip neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 2
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Lung adenocarcinoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 9 | 4
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 5 | 8
Lung squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 4 | 4
Malignant neoplasm of renal pelvis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Malignant neoplasm of uterine adnexa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Malignant peritoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Mesothelioma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Metastases to bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Metastases to bone marrow (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Metastatic bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 4 | 1
Metastatic carcinoma of the bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3 | 1
Metastatic gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3 | 6
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 3
Metastatic uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 6 | 2
Mycosis fungoides (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Neoplasm of appendix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Neoplasm prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Neurilemmoma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Neuroectodermal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 2
Non-Hodgkin's lymphoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3 | 1
Non-small cell lung cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Esophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1
Esophageal squamous cell carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Oligodendroglioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Oral papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Ovarian granulosa-theca cell tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Pancoast's tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3 | 3
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 5 | 5
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Parathyroid tumor benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Pituitary tumor benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 2
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Porocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 26 | 20
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 7 | 4
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Prostate cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Prostate cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 6 | 5
Rectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 6 | 5
Rectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 2
Rectosigmoid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3 | 1
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Renal cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 4
Renal cell carcinoma stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Rhabdomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Salivary gland adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Salivary gland cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Sarcoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3 | 0
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 2
Spinal hemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Superficial spreading melanoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Teratoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 5 | 0
Ureteric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Ureteric cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 4 | 2
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3 | 0
Vulval cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Amnesia (Nervous system disorders) | 0 | 0 | 1
Apallic syndrome (Nervous system disorders) | 0 | 0 | 1
Basal ganglia hemorrhage (Nervous system disorders) | 0 | 0 | 1
Basilar artery stenosis (Nervous system disorders) | 0 | 1 | 0
Brain injury (Nervous system disorders) | 0 | 1 | 0
Brain stem hemorrhage (Nervous system disorders) | 0 | 0 | 1
Brain stem infarction (Nervous system disorders) | 0 | 1 | 2
Brain stem stroke (Nervous system disorders) | 0 | 1 | 0
Carotid arteriosclerosis (Nervous system disorders) | 0 | 0 | 1
Carotid artery occlusion (Nervous system disorders) | 0 | 0 | 2
Carotid artery stenosis (Nervous system disorders) | 2 | 30 | 32
Carotid sinus syndrome (Nervous system disorders) | 0 | 0 | 1
Carpal tunnel syndrome (Nervous system disorders) | 2 | 9 | 6
Central nervous system lesion (Nervous system disorders) | 0 | 1 | 0
Cerebellar infarction (Nervous system disorders) | 0 | 1 | 3
Cerebellar ischemia (Nervous system disorders) | 0 | 1 | 0
Cerebellar syndrome (Nervous system disorders) | 0 | 2 | 1
Cerebral artery embolism (Nervous system disorders) | 0 | 0 | 1
Cerebral artery stenosis (Nervous system disorders) | 0 | 0 | 1
Cerebral cyst (Nervous system disorders) | 0 | 1 | 0
Cerebral hematoma (Nervous system disorders) | 0 | 2 | 0
Cerebral hemorrhage (Nervous system disorders) | 0 | 2 | 2
Cerebral infarction (Nervous system disorders) | 2 | 15 | 12
Cerebral ischemia (Nervous system disorders) | 0 | 3 | 7
Cerebral thrombosis (Nervous system disorders) | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 8 | 46 | 44
Cerebrovascular insufficiency (Nervous system disorders) | 0 | 0 | 1
Cervical myelopathy (Nervous system disorders) | 1 | 1 | 1
Cervicobrachial syndrome (Nervous system disorders) | 0 | 2 | 1
Cluster headache (Nervous system disorders) | 0 | 0 | 1
Cognitive disorder (Nervous system disorders) | 0 | 0 | 1
Coma (Nervous system disorders) | 0 | 1 | 0
Complicated migraine (Nervous system disorders) | 0 | 0 | 1
Cubital tunnel syndrome (Nervous system disorders) | 0 | 0 | 1
Dementia (Nervous system disorders) | 0 | 1 | 0
Dementia Alzheimer's type (Nervous system disorders) | 0 | 1 | 0
Diabetic encephalopathy (Nervous system disorders) | 0 | 1 | 0
Diabetic neuropathy (Nervous system disorders) | 1 | 6 | 8
Dizziness (Nervous system disorders) | 1 | 2 | 6
Dysaesthesia (Nervous system disorders) | 1 | 0 | 0
Dysarthria (Nervous system disorders) | 0 | 1 | 2
Dysstasia (Nervous system disorders) | 0 | 1 | 0
Embolic stroke (Nervous system disorders) | 0 | 1 | 2
Encephalopathy (Nervous system disorders) | 0 | 0 | 1
Epidural lipomatosis (Nervous system disorders) | 0 | 1 | 0
Epilepsy (Nervous system disorders) | 1 | 3 | 1
Facial palsy (Nervous system disorders) | 0 | 3 | 1
Facial paresis (Nervous system disorders) | 0 | 1 | 1
Hemorrhage intracranial (Nervous system disorders) | 1 | 1 | 1
Hemorrhagic stroke (Nervous system disorders) | 2 | 6 | 3
Hemorrhagic transformation stroke (Nervous system disorders) | 0 | 0 | 1
Head titubation (Nervous system disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 2 | 4 | 6
Hemiparesis (Nervous system disorders) | 0 | 1 | 2
Hepatic encephalopathy (Nervous system disorders) | 0 | 1 | 0
Hypertensive encephalopathy (Nervous system disorders) | 0 | 0 | 1
Hypoglycemic coma (Nervous system disorders) | 0 | 0 | 1
Hypoxic encephalopathy (Nervous system disorders) | 0 | 2 | 1
IIIrd nerve paresis (Nervous system disorders) | 0 | 1 | 0
Incoherent (Nervous system disorders) | 0 | 1 | 1
Intercostal neuralgia (Nervous system disorders) | 0 | 0 | 1
Intracranial aneurysm (Nervous system disorders) | 0 | 1 | 0
Intracranial hematoma (Nervous system disorders) | 0 | 1 | 0
Ischemic cerebral infarction (Nervous system disorders) | 0 | 2 | 1
Ischemic stroke (Nervous system disorders) | 2 | 42 | 22
IVth nerve paresis (Nervous system disorders) | 0 | 0 | 1
Lacunar infarction (Nervous system disorders) | 0 | 1 | 6
Lethargy (Nervous system disorders) | 0 | 0 | 1
Loss of consciousness (Nervous system disorders) | 0 | 7 | 6
Lumbar radiculopathy (Nervous system disorders) | 0 | 2 | 1
Meralgia paraesthetica (Nervous system disorders) | 0 | 0 | 1
Metabolic encephalopathy (Nervous system disorders) | 0 | 1 | 0
Migraine (Nervous system disorders) | 0 | 2 | 1
Migraine with aura (Nervous system disorders) | 0 | 0 | 1
Myasthenia gravis (Nervous system disorders) | 0 | 1 | 0
Myelitis transverse (Nervous system disorders) | 0 | 0 | 1
Myelopathy (Nervous system disorders) | 1 | 0 | 0
Nerve compression (Nervous system disorders) | 1 | 4 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 2
Paraesthesia (Nervous system disorders) | 0 | 1 | 2
Paralysis (Nervous system disorders) | 0 | 0 | 1
Parkinson's disease (Nervous system disorders) | 0 | 1 | 2
Parkinsonism (Nervous system disorders) | 0 | 0 | 1
Polyneuropathy (Nervous system disorders) | 0 | 2 | 3
Post-herpetic neuralgia (Nervous system disorders) | 0 | 1 | 0
Post-traumatic epilepsy (Nervous system disorders) | 0 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 7 | 7
Pseudoradicular syndrome (Nervous system disorders) | 0 | 1 | 0
Radial nerve palsy (Nervous system disorders) | 0 | 1 | 0
Radicular pain (Nervous system disorders) | 0 | 1 | 0
Radicular syndrome (Nervous system disorders) | 0 | 2 | 0
Radiculopathy (Nervous system disorders) | 0 | 1 | 1
Reversible ischemic neurological deficit (Nervous system disorders) | 0 | 0 | 1
Sciatica (Nervous system disorders) | 1 | 8 | 4
Somnolence (Nervous system disorders) | 0 | 0 | 2
Spinal claudication (Nervous system disorders) | 0 | 1 | 0
Spinal cord infarction (Nervous system disorders) | 0 | 1 | 1
Spondylitic myelopathy (Nervous system disorders) | 0 | 1 | 0
Subarachnoid hemorrhage (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 2 | 19 | 21
Thalamic infarction (Nervous system disorders) | 0 | 0 | 1
Transient global amnesia (Nervous system disorders) | 0 | 0 | 2
Transient ischemic attack (Nervous system disorders) | 3 | 34 | 36
Tremor (Nervous system disorders) | 0 | 1 | 1
Trigeminal neuralgia (Nervous system disorders) | 0 | 2 | 1
Vascular dementia (Nervous system disorders) | 0 | 1 | 1
Vascular encephalopathy (Nervous system disorders) | 0 | 1 | 1
Vertebral artery occlusion (Nervous system disorders) | 0 | 0 | 1
Vertebral artery stenosis (Nervous system disorders) | 0 | 2 | 1
Vertebrobasilar insufficiency (Nervous system disorders) | 2 | 5 | 8
Vertigo CNS origin (Nervous system disorders) | 0 | 0 | 2
VIIth nerve paralysis (Nervous system disorders) | 1 | 0 | 0
VIth nerve paralysis (Nervous system disorders) | 0 | 0 | 1
Abnormal behavior (Psychiatric disorders) | 0 | 1 | 0
Acute psychosis (Psychiatric disorders) | 0 | 1 | 0
Adjustment disorder (Psychiatric disorders) | 0 | 0 | 1
Alcoholism (Psychiatric disorders) | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1 | 0
Bereavement reaction (Psychiatric disorders) | 0 | 1 | 0
Completed suicide (Psychiatric disorders) | 0 | 1 | 1
Confusional state (Psychiatric disorders) | 0 | 5 | 3
Conversion disorder (Psychiatric disorders) | 0 | 2 | 0
Delirium (Psychiatric disorders) | 0 | 2 | 0
Depression (Psychiatric disorders) | 0 | 3 | 10
Hallucination, visual (Psychiatric disorders) | 0 | 1 | 0
Hypochondriasis (Psychiatric disorders) | 0 | 1 | 0
Mood disorder due to a general medical condition (Psychiatric disorders) | 0 | 0 | 2
Personality disorder (Psychiatric disorders) | 0 | 1 | 0
Post-traumatic stress disorder (Psychiatric disorders) | 0 | 1 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 1 | 0
Schizoaffective disorder (Psychiatric disorders) | 0 | 0 | 1
Schizophreniform disorder (Psychiatric disorders) | 0 | 1 | 0
Suicide attempt (Psychiatric disorders) | 0 | 0 | 1
Acute prerenal failure (Renal and urinary disorders) | 0 | 1 | 0
Azotemia (Renal and urinary disorders) | 0 | 2 | 1
Bladder neck obstruction (Renal and urinary disorders) | 1 | 1 | 0
Bladder neck sclerosis (Renal and urinary disorders) | 0 | 0 | 1
Bladder obstruction (Renal and urinary disorders) | 0 | 1 | 0
Bladder prolapse (Renal and urinary disorders) | 0 | 1 | 1
Bladder stenosis (Renal and urinary disorders) | 0 | 0 | 1
Bladder tamponade (Renal and urinary disorders) | 0 | 1 | 0
Calculus bladder (Renal and urinary disorders) | 1 | 0 | 1
Calculus ureteric (Renal and urinary disorders) | 0 | 6 | 2
Calculus urethral (Renal and urinary disorders) | 0 | 0 | 1
Calculus urinary (Renal and urinary disorders) | 0 | 1 | 2
Cystitis hemorrhagic (Renal and urinary disorders) | 1 | 2 | 1
Diabetic nephropathy (Renal and urinary disorders) | 0 | 2 | 1
Hematuria (Renal and urinary disorders) | 1 | 6 | 4
Hydronephrosis (Renal and urinary disorders) | 0 | 4 | 1
Nephrolithiasis (Renal and urinary disorders) | 2 | 13 | 11
Nephropathy (Renal and urinary disorders) | 0 | 1 | 0
Nephropathy toxic (Renal and urinary disorders) | 0 | 0 | 1
Nephrotic syndrome (Renal and urinary disorders) | 0 | 2 | 1
Obstructive uropathy (Renal and urinary disorders) | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1
Pyuria (Renal and urinary disorders) | 0 | 1 | 0
Renal artery arteriosclerosis (Renal and urinary disorders) | 0 | 1 | 0
Renal artery stenosis (Renal and urinary disorders) | 0 | 4 | 6
Renal artery thrombosis (Renal and urinary disorders) | 0 | 1 | 0
Renal colic (Renal and urinary disorders) | 0 | 5 | 2
Renal cyst (Renal and urinary disorders) | 0 | 0 | 1
Renal disorder (Renal and urinary disorders) | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 3 | 17 | 18
Renal failure acute (Renal and urinary disorders) | 5 | 18 | 15
Renal failure chronic (Renal and urinary disorders) | 0 | 9 | 11
Renal hypertension (Renal and urinary disorders) | 0 | 0 | 1
Renal impairment (Renal and urinary disorders) | 0 | 4 | 4
Renal tubular necrosis (Renal and urinary disorders) | 0 | 1 | 0
Stress urinary incontinence (Renal and urinary disorders) | 0 | 4 | 1
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 | 1 | 1
Ureteric obstruction (Renal and urinary disorders) | 0 | 0 | 1
Ureteric stenosis (Renal and urinary disorders) | 0 | 2 | 0
Urethral caruncle (Renal and urinary disorders) | 0 | 1 | 0
Urethral hemorrhage (Renal and urinary disorders) | 1 | 0 | 0
Urethral meatus stenosis (Renal and urinary disorders) | 0 | 5 | 0
Urethral stenosis (Renal and urinary disorders) | 1 | 5 | 5
Urinary bladder hemorrhage (Renal and urinary disorders) | 0 | 1 | 0
Urinary bladder polyp (Renal and urinary disorders) | 0 | 1 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 2 | 2
Urinary retention (Renal and urinary disorders) | 2 | 3 | 2
Urinary tract obstruction (Renal and urinary disorders) | 2 | 2 | 1
Acquired hydrocele (Reproductive system and breast disorders) | 0 | 0 | 1
Adenomyosis (Reproductive system and breast disorders) | 0 | 1 | 0
Balanitis (Reproductive system and breast disorders) | 0 | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 8 | 39 | 30
Breast hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 1
Breast mass (Reproductive system and breast disorders) | 0 | 1 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 0 | 1
Cervical polyp (Reproductive system and breast disorders) | 0 | 1 | 0
Colpocele (Reproductive system and breast disorders) | 0 | 2 | 1
Cystocele (Reproductive system and breast disorders) | 0 | 2 | 0
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 | 3 | 1
Endometrial hypertrophy (Reproductive system and breast disorders) | 0 | 1 | 0
Epididymal cyst (Reproductive system and breast disorders) | 0 | 1 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 1
Fibrocystic breast disease (Reproductive system and breast disorders) | 0 | 1 | 0
Genital prolapse (Reproductive system and breast disorders) | 0 | 0 | 1
Gynecomastia (Reproductive system and breast disorders) | 0 | 0 | 1
Metrorrhagia (Reproductive system and breast disorders) | 0 | 1 | 1
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0 | 2
Ovarian cyst torsion (Reproductive system and breast disorders) | 1 | 0 | 1
Posthitis (Reproductive system and breast disorders) | 0 | 1 | 0
Prostatism (Reproductive system and breast disorders) | 0 | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 1 | 4 | 0
Prostatomegaly (Reproductive system and breast disorders) | 0 | 1 | 1
Rectocele (Reproductive system and breast disorders) | 0 | 0 | 2
Scrotal cyst (Reproductive system and breast disorders) | 0 | 1 | 0
Testicular swelling (Reproductive system and breast disorders) | 0 | 1 | 0
Uterine polyp (Reproductive system and breast disorders) | 1 | 3 | 3
Uterine prolapse (Reproductive system and breast disorders) | 1 | 3 | 5
Uterovaginal prolapse (Reproductive system and breast disorders) | 0 | 0 | 1
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0
Vaginal prolapse (Reproductive system and breast disorders) | 1 | 0 | 3
Acute pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 | 7 | 9
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 5
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 12 | 7
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Brain hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Bronchial dysplasia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Choking (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 6 | 17 | 21
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 18 | 18
Dyspnea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 5 | 3
Foreign body aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Hemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 4
Laryngeal granuloma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasal septum perforation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Nasal turbinate hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Organizing pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pickwickian syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 5 | 7
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 4
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 3
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 15 | 11
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 2
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 | 15 | 13
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 9
Restrictive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Sleep apnea syndrome (Respiratory, thoracic and mediastinal disorders) | 3 | 14 | 14
Snoring (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Upper airway obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Vocal cord inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1 | 4
Cold sweat (Skin and subcutaneous tissue disorders) | 0 | 2 | 3
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Diabetic bullosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Diabetic neuropathic ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Diabetic ulcer (Skin and subcutaneous tissue disorders) | 1 | 2 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dry gangrene (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Erythema nodosum (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hidradenitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Hirsutism (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 3 | 4
Hypoaesthesia facial (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Leukocytoclastic vasculitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Lichen sclerosis (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Necrobiosis lipoidica diabeticorum (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Neuropathic ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Psoriasis (Skin and subcutaneous tissue disorders) | 2 | 2 | 1
Pyoderma gangrenosum (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Scar pain (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Sebaceous hyperplasia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 5 | 5
Activities of daily living impaired (Social circumstances) | 0 | 1 | 0
Family stress (Social circumstances) | 0 | 0 | 1
Social stay hospitalization (Social circumstances) | 0 | 1 | 1
Cardiac pacemaker battery replacement (Surgical and medical procedures) | 0 | 0 | 2
Cardiac pacemaker replacement (Surgical and medical procedures) | 0 | 3 | 3
Cholecystectomy (Surgical and medical procedures) | 0 | 0 | 1
Coronary artery bypass (Surgical and medical procedures) | 0 | 0 | 1
Diabetes mellitus management (Surgical and medical procedures) | 0 | 2 | 1
Drug therapy changed (Surgical and medical procedures) | 0 | 1 | 0
Gastric banding (Surgical and medical procedures) | 0 | 1 | 0
Hip arthroplasty (Surgical and medical procedures) | 0 | 0 | 1
Hysterectomy (Surgical and medical procedures) | 0 | 1 | 0
Implantable defibrillator replacement (Surgical and medical procedures) | 0 | 3 | 1
Intra-uterine contraceptive device removal (Surgical and medical procedures) | 0 | 1 | 0
Liposuction (Surgical and medical procedures) | 0 | 0 | 1
Medical device change (Surgical and medical procedures) | 0 | 1 | 0
Rehabilitation therapy (Surgical and medical procedures) | 0 | 0 | 1
Therapeutic procedure (Surgical and medical procedures) | 0 | 1 | 1
Accelerated hypertension (Vascular disorders) | 0 | 4 | 3
Angiodysplasia (Vascular disorders) | 0 | 1 | 0
Aortic aneurysm (Vascular disorders) | 1 | 12 | 13
Aortic aneurysm rupture (Vascular disorders) | 0 | 1 | 5
Aortic arteriosclerosis (Vascular disorders) | 0 | 1 | 0
Aortic dilatation (Vascular disorders) | 0 | 0 | 1
Aortic dissection (Vascular disorders) | 0 | 2 | 1
Aortic rupture (Vascular disorders) | 0 | 0 | 1
Aortic stenosis (Vascular disorders) | 0 | 7 | 3
Arterial disorder (Vascular disorders) | 0 | 4 | 1
Arterial insufficiency (Vascular disorders) | 0 | 1 | 0
Arterial occlusive disease (Vascular disorders) | 1 | 1 | 0
Arterial rupture (Vascular disorders) | 0 | 0 | 1
Arterial stenosis (Vascular disorders) | 1 | 0 | 1
Arterial stenosis limb (Vascular disorders) | 0 | 6 | 6
Arterial thrombosis (Vascular disorders) | 0 | 1 | 0
Arterial thrombosis limb (Vascular disorders) | 0 | 1 | 0
Arteriosclerosis (Vascular disorders) | 0 | 4 | 2
Arteriosclerosis obliterans (Vascular disorders) | 0 | 6 | 2
Arteriovenous fistula (Vascular disorders) | 1 | 0 | 2
Arteritis (Vascular disorders) | 1 | 2 | 1
Circulatory collapse (Vascular disorders) | 2 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 13 | 15
Diabetic microangiopathy (Vascular disorders) | 0 | 0 | 1
Diabetic vascular disorder (Vascular disorders) | 0 | 1 | 0
Embolism (Vascular disorders) | 0 | 1 | 0
Exsanguination (Vascular disorders) | 0 | 0 | 1
Extremity necrosis (Vascular disorders) | 1 | 3 | 2
Femoral arterial stenosis (Vascular disorders) | 2 | 18 | 13
Femoral artery aneurysm (Vascular disorders) | 0 | 1 | 1
Femoral artery occlusion (Vascular disorders) | 0 | 10 | 8
Hematoma (Vascular disorders) | 0 | 4 | 1
Hemorrhage (Vascular disorders) | 0 | 1 | 0
Hot flush (Vascular disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 2 | 17 | 26
Hypertensive crisis (Vascular disorders) | 0 | 5 | 10
Hypertensive emergency (Vascular disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 1 | 2 | 5
Iliac artery occlusion (Vascular disorders) | 0 | 2 | 2
Iliac artery stenosis (Vascular disorders) | 0 | 6 | 3
Intermittent claudication (Vascular disorders) | 2 | 4 | 1
Lymphedema (Vascular disorders) | 0 | 2 | 2
Macroangiopathy (Vascular disorders) | 0 | 1 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 4 | 3
Pallor (Vascular disorders) | 0 | 1 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 3 | 52 | 39
Peripheral artery aneurysm (Vascular disorders) | 1 | 1 | 6
Peripheral embolism (Vascular disorders) | 0 | 4 | 4
Peripheral ischemia (Vascular disorders) | 1 | 16 | 14
Peripheral vascular disorder (Vascular disorders) | 0 | 12 | 11
Phlebitis (Vascular disorders) | 0 | 1 | 0
Phlebitis superficial (Vascular disorders) | 0 | 1 | 0
Post thrombotic syndrome (Vascular disorders) | 0 | 1 | 0
Shock (Vascular disorders) | 0 | 1 | 0
Shock hemorrhagic (Vascular disorders) | 1 | 4 | 3
Subclavian artery stenosis (Vascular disorders) | 0 | 1 | 0
Subclavian artery thrombosis (Vascular disorders) | 0 | 1 | 0
Subclavian steal syndrome (Vascular disorders) | 1 | 0 | 1
Subclavian vein thrombosis (Vascular disorders) | 0 | 1 | 0
Temporal arteritis (Vascular disorders) | 0 | 0 | 2
Thromboangiitis obliterans (Vascular disorders) | 0 | 1 | 0
Thrombophlebitis (Vascular disorders) | 0 | 2 | 1
Thrombophlebitis superficial (Vascular disorders) | 0 | 0 | 2
Thrombosis (Vascular disorders) | 0 | 0 | 2
Varicophlebitis (Vascular disorders) | 0 | 1 | 0
Varicose ulceration (Vascular disorders) | 0 | 1 | 1
Varicose vein (Vascular disorders) | 1 | 14 | 2
Vascular rupture (Vascular disorders) | 0 | 0 | 1
Vascular shunt (Vascular disorders) | 0 | 0 | 1
Vascular stenosis (Vascular disorders) | 0 | 1 | 1
Vasculitis (Vascular disorders) | 0 | 0 | 1
Vasculitis necrotizing (Vascular disorders) | 0 | 1 | 0
Venous insufficiency (Vascular disorders) | 0 | 8 | 3
Venous thrombosis (Vascular disorders) | 1 | 1 | 0
Venous thrombosis limb (Vascular disorders) | 0 | 1 | 2

LIMITATIONS AND CAVEATS:
Most subjects not indicated for sibutramine (sbt) due to CV disease. Long-term sbt use (6 yrs) regardless of weight loss, is inconsistent with label (limits use to 1-2 yrs & 5% weight loss). Trial lacked true placebo; all received Lead-in Period sbt.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Abbott requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. Abbott requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if Abbott needs to secure patent or proprietary protection.